CLINICAL TRIAL: NCT00970749
Title: Antigen-specific Cell Mediated Immune Response to Chlamydia Trachomatis
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: PRO09070184; U19AI084024 (NIH)
Record Dates: First submitted 2009-08-29; First posted 2009-09-02 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Chlamydia
Keywords: chlamydia; healthy women; history of endocervical chlamydia; no history of endocervical chlamydia
MeSH Terms: conditions — Chlamydia Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- history of chlamydia infection: Women who self-reported a history of cervical infection with Chlamydia trachomatis
- no history of chlamydia infection: Women who self-reported no history of cervical infection with Chlamydia trachomatis

SUMMARY:
This is an exploratory study in which the investigators will develop a way to identify the cell responses most strongly associated with protection against chlamydia infection. This study is not driven by a hypothesis.

DETAILED DESCRIPTION:
With more than 90 million new cases annually, Chlamydia trachomatis is the most common sexually transmitted bacterial disease. Untreated endocervical C. trachomatis infections can cause pelvic inflammatory disease (PID), a disorder of the endometrium, fallopian tubes, and adjacent structures that occurs after ascension of the bacterium from the lower to upper genital tract. Adverse outcomes secondary to C. trachomatis-induced PID include tubal infertility, ectopic pregnancy, and chronic pelvic pain. Vaccine development has been identified as essential for control of C. trachomatis infections, and current evidence suggests that an effective vaccine will likely be based on several C. trachomatis antigens. Experimental models of infection have identified HSP60, major outer-membrane protein (MOMP), outer membrane protein 2 (OMP2), and polymorphic membrane protein D (PmpD) as promising vaccine candidates. A prospective study of Kenyan commercial sex workers found that production of interferon-gamma (IFN-γ) by peripheral blood cells stimulated with chlamydia heat-shock protein (HSP60) strongly correlated with protection against incident C. trachomatis infection. This proposal details an exploratory identification of the antigen-specific cell mediated immune responses associated with antecedent C. trachomatis infection in women.

C. trachomatis is an obligate, intracellular, gram-negative microorganism recognized as the most common bacterial sexually transmitted disease worldwide. The highest rates of infection with this organism are consistently found among adolescents and young adults. Young women are also the group most adversely impacted by the effects of C. trachomatis infection on reproductive health. While approximately 70% of infections with C. trachomatis in young women are asymptomatic, 20% - 40% of these occult infections will progress from endocervical inflammation to the development of PID. In addition to its strong association with PID, C. trachomatis infection is also thought to enhance HIV transmission and contribute to human papilloma virus induced cervical neoplasia. Although data from both experimental models and clinical studies suggest that antigen specific CD4+ and CD8+ T cells are required for optimal control of genital tract chlamydial infections, the current lack of information regarding the specific C. trachomatis antigens eliciting protective immune responses in humans hinders vaccine development.

This is an exploratory investigation in which we will develop the methodology needed to identify the antigen-specific cell mediated immune responses most strongly associated with protection against incident C. trachomatis infection.

ELIGIBILITY:
Inclusion Criteria:

* Women between 15-35 years of age at the time of enrollment onto this study. Minors between the ages of 1-17 will require parental consent to participate in the study.
* History of, in past 5 years, endocervical C. trachomatis infection (total of 20 women) or no history of endocervical C. trachomatis infection (total of 10 women).

Exclusion Criteria:

* Pregnancy.
* Immunocompromised, by history (including but not limited to known HIV, cancer, autoimmune diseases).

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 20 women with history of endocervical chlamydia and 10 women with no history of endocervical chlamydia
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
This is an exploratory investigation in which we will develop the methodology needed to identify the antigen-specific cell mediated immune responses most strongly associated with protection against incident C. trachomatis infection. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Cherpes, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No